CLINICAL TRIAL: NCT00545935
Title: Safety and Efficacy of Methylene Blue Combined With Amodiaquine or Artesunate for Malaria Treatment in Children of Burkina Faso: RCT in the Frame of the A8 Project of SFB 544
Brief Title: Safety and Efficacy of Methylene Blue Combined With Amodiaquine or Artesunate for Malaria Treatment in Children of Burkina Faso
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB-2007b
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination

ARMS (3):
- 1-Methylenblue-Amodiaquine (Active Comparator)
  Interventions: Drug: Methylenblue-Amodiaquine (MB-AQ)
- 2-Methylenblue-Artesunate (Active Comparator)
  Interventions: Drug: Methylenblue-Artesunate (MB-AS)
- 3-Artesunate-Amodiaquine (Active Comparator)
  Interventions: Drug: Artesunate-Amodiaquine (AS-AQ)

INTERVENTIONS:
Drug: Methylenblue-Amodiaquine (MB-AQ) — For 3 days twice daily 10 mg/kg MB accompanied by once daily 10 mg/kg AQ
  Arms: 1-Methylenblue-Amodiaquine
Drug: Methylenblue-Artesunate (MB-AS) — 3 days once daily 4 mg/kg AS accompanied by twice daily 10 mg/kg MB given over 7 days
  Arms: 2-Methylenblue-Artesunate
Drug: Artesunate-Amodiaquine (AS-AQ) — For 3 days once daily 10 mg/kg AQ accompanied by 4mg/kg AS.
  Arms: 3-Artesunate-Amodiaquine

SUMMARY:
The purpose of the study is to investigate the safety and efficacy profile of a new paediatric MB formulation combined with AQ or AS and compared to AS-AQ in young African children with uncomplicated falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* 0.5-5 year (6-59 months) old children
* uncomplicated malaria caused by P. falciparum
* asexual parasites ≥ 2000/µ and ≤ 200000/µ
* axillary temperature ≥ 37.5 Celsius or a history of fever during last 24 hours
* Burkinabe nationality
* informed consent

Exclusion Criteria:

* complicated or severe malaria
* any apparent significant disease
* anaemia (haematocrit < 21%)
* treated in the same trial before
* modern antimalarial treatment prior to inclusion (last three days), except children having been treated with chloroquine

Ages: 6 Months to 59 Months | Sex: All
Age Groups: Child
Enrollment: 186
Dates: Start 2007-07; Study Completion 2007-10

PRIMARY OUTCOMES:
Incidence of observed and self-reported non-serious adverse events over the 28 days observation period | 28 days

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAE) and the adequate clinical and parasitological response rate (ACPR) | 28 days
Early treatment failure (ETF) rate | 28 days
Late clinical failure (LCF) rate at D14 and D28 | 28 days
Late parasitological failure (LPF) rate at D14 and D28 | 28 days
Fever clearance time | 28 days
Parasite clearance time | 28 days
Change in haematocrit after 2,14 and 28 days compared to baseline | 28 days
MB whole blood concentrations on D3,5 or 7 compared to concentrations after the first dose | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Mueller, Prof., Principal Investigator — Heidelberg University
Locations (1):
- Centre de Recherche en Sante de Nouna, Nouna, Burkina Faso